CLINICAL TRIAL: NCT03331783
Title: The Evaluation of the Effect of Output on Newly Developed Adhesives
Brief Title: Assessment of the Effect of Output on New Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_21_22
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Ileostomy - Stoma
MeSH Terms: interventions — cholecystokinin 33 (10-20)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of new adhesive strips (Experimental): On the peristomal skin 4 different patches are applied to the skin (Standard hydrocolloid adhesive patch; LT-2, LT21 and 33-20. There is a bag welded to each patch. Tthe bag contains real output.
  The difference between the four patches is that they are made of four different adhesives.
  The primary endpoint is measured after 8 hours and 24 hours.
  Interventions: Other: Standard hydrocolloid adhesive patch; Other: LT-2; Other: LT-21; Other: 33-20

INTERVENTIONS:
Other: Standard hydrocolloid adhesive patch — This patch is made of a standard hydrocolloid adhesive
Other: LT-2 — This patch is made of a new adhesive
Other: LT-21 — This patch is made of a new adhesive
Other: 33-20 — This patch is made of a new adhesive

SUMMARY:
The study investigates the impact real output has on adhesion of new adhesives

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have had a stoma for more than one year
* Have intact skin on the area used in the evaluation
* Has a stoma with a diameter up to (≤) 35 mm
* Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

* Currently receiving or have within the past 2 month received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
* Are pregnant or breastfeeding
* Having dermatological problems in the peri-stomal- or abdominal area (assessed by investigating scientist)
* Actively participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 8 hours
  The trans epidermal water loss is measured on the peristomal skin using a probe. The trans epidermal water loss is a measure for the skins barrier function. There is always a loss of water from the skin due to natural evaporation. However, when the skin barrier is damaged the evaporation will increase leading to an increase in the trans epidermal water loss.Thus, trans epidermal water loss is used to assess the damage to the skin. Maesurents are taken at time 0 and after 8 hours of output exposure to the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Feldskov, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark